CLINICAL TRIAL: NCT03312192
Title: Stand-Alone Cage Versus Anterior Plating for 1-2 Level Anterior Cervical Discectomy and Fusion. A Clinical and Radiographic Analysis
Brief Title: Stand-Alone Cage Verus Anterior Plating for Anterior Cervical Discectomy and Fusion.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Carla Edwards, Clinical Research Manger, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14021901
Record Dates: First submitted 2017-08-08; First posted 2017-10-17 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Degenerative Disc Disease; Cervical Spine Degeneration
Keywords: Anterior Cervical Discectomy and Fusion; Stand-Alone Cage; Anterior Plating
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: 1. Stand-alone ACDF, which means the placement of an interbody device (cage) without anterior fixation or plating; 2. ACDF with and interbody cage and anterior plating for fixation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Plate and Cage (Active Comparator): ACDF with interbody cage and anterior plating.
  Interventions: Device: Interbody Cage and Anterior Plating
- Stand Alone Cage (Active Comparator): ACDF with stand alone interbody cage without anterior plating
  Interventions: Device: Interbody Cage

INTERVENTIONS:
Device: Interbody Cage — Anterior cervical discectomy and fusion with interbody cage placement
  Arms: Stand Alone Cage
Device: Interbody Cage and Anterior Plating — Anterior cervical discectomy and fusion with interbody cage placement and anterior plating
  Arms: Plate and Cage

SUMMARY:
The purpose of this study is to compare the clinical results between two different techniques for ACDF: 1. Stand-alone ACDF, which means the placement of an interbody device (cage) without anterior fixation or plating; 2. ACDF with and interbody cage and anterior plating for fixation. Both of these procedures are commonly performed at Rush with unclear advantage of one procedure over the other. Both have been associated with good to excellent clinical outcomes. The devices used in this study are approved by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
Anterior cervical discectomy and fusion (ACDF) is one the most common procedures performed by spine surgeons. Although ACDF with autologous bone graft and anterior plating is commonly performed, this procedure may be associated with postoperative dysphagia, significant costs and adjacent segment pathology. To address these concerns, a number of surgeons have opted to utilize an interbody cage in a stand-alone fashion with good to excellent results. However, the published data is limited and currently there in no consensus among spine surgeons regarding the best technique to achieve fusion and improve clinical outcomes in patients with degenerative disc disease in the cervical spine.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary 1- to 2-level ACDF

  (a) Diagnosis: myelopathy, radiculopathy, myeloradiculopathy, stenosis, herniated nucleus pulposus, degenerative disc disease, spondylosis, osteophytic complexes, and foraminal stenosis
* Patients able to provide informed consent

Exclusion Criteria:

* Cervical spine trauma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement - Change in Baseline Visual analogue Score (VAS) for Pain | 6 months
  Patients will be asked to complete the VAS to measure their pain prior to surgery and at their preoperative office visit(s) or just prior to surgery in the preoperative waiting area. Scores at the 6 month follow up office visit will be compared to baseline

SECONDARY OUTCOMES:
Dysphagia | 6 months
  6 month postoperative followup SWAL-QOL score will be compared to baseline
Fusion Rates | 6 months
  Postoperative radiographic studies will be performed at 6 month follow up visit to assess for arthrodesis (fusion) and pseudarthrosis (non-fusion).
Clinical Improvement - Change in baseline 12-item Short Form (SF-12) Health Survey at 6 months | 6 months
  SF-12 survey scores at 6 month follow up will be compared to baseline
Clinical Improvement - Change in baseline Oswestry Disability Index (ODI) at 6 months | 6 months
  ODI survey scores at 6 month follow up will be compared to baseline

OTHER OUTCOMES:
Adverse Events | 1 year
  (a) Intra-operative - Information will be obtained from the operative note. (i) Blood loss, length of surgery, procedural details, complications (b) Post-operative - Information will be obtained from the clinic notes
Narcotics Consumption | 3 days
  The total amount of narcotic use for each subject will be recorded. Dosages of narcotics will be converted to morphine equivalents. This information will be measured during the hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Kern Singh, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ji GY, Oh CH, Shin DA, Ha Y, Kim KN, Yoon DH, Yudoyono F. Stand-alone Cervical Cages Versus Anterior Cervical Plates in 2-Level Cervical Anterior Interbody Fusion Patients: Analysis of Adjacent Segment Degeneration. J Spinal Disord Tech. 2015 Aug;28(7):E433-8. doi: 10.1097/BSD.0b013e3182a355ad. PMID 23897053
- [Background] Choi KC, Ryu KS, Lee SH, Kim YH, Lee SJ, Park CK. Biomechanical comparison of anterior lumbar interbody fusion: stand-alone interbody cage versus interbody cage with pedicle screw fixation -- a finite element analysis. BMC Musculoskelet Disord. 2013 Jul 26;14:220. doi: 10.1186/1471-2474-14-220. PMID 23890389
- [Background] Oh JK, Kim TY, Lee HS, You NK, Choi GH, Yi S, Ha Y, Kim KN, Yoon DH, Shin HC. Stand-alone cervical cages versus anterior cervical plate in 2-level cervical anterior interbody fusion patients: clinical outcomes and radiologic changes. J Spinal Disord Tech. 2013 Dec;26(8):415-20. doi: 10.1097/BSD.0b013e31824c7d22. PMID 22367466
- [Background] Lee MJ, Dettori JR, Standaert CJ, Ely CG, Chapman JR. Indication for spinal fusion and the risk of adjacent segment pathology: does reason for fusion affect risk? A systematic review. Spine (Phila Pa 1976). 2012 Oct 15;37(22 Suppl):S40-51. doi: 10.1097/BRS.0b013e31826ca9b1. PMID 22872219
- [Background] Hilibrand AS, Robbins M. Adjacent segment degeneration and adjacent segment disease: the consequences of spinal fusion? Spine J. 2004 Nov-Dec;4(6 Suppl):190S-194S. doi: 10.1016/j.spinee.2004.07.007. PMID 15541666
- [Background] Cho SK, Riew KD. Adjacent segment disease following cervical spine surgery. J Am Acad Orthop Surg. 2013 Jan;21(1):3-11. doi: 10.5435/JAAOS-21-01-3. PMID 23281466
- [Background] Kraemer P, Fehlings MG, Hashimoto R, Lee MJ, Anderson PA, Chapman JR, Raich A, Norvell DC. A systematic review of definitions and classification systems of adjacent segment pathology. Spine (Phila Pa 1976). 2012 Oct 15;37(22 Suppl):S31-9. doi: 10.1097/BRS.0b013e31826d7dd6. PMID 22885835
- [Background] Mobbs RJ, Rao P, Chandran NK. Anterior cervical discectomy and fusion: analysis of surgical outcome with and without plating. J Clin Neurosci. 2007 Jul;14(7):639-42. doi: 10.1016/j.jocn.2006.04.003. PMID 17532499
- [Background] Savolainen S, Rinne J, Hernesniemi J. A prospective randomized study of anterior single-level cervical disc operations with long-term follow-up: surgical fusion is unnecessary. Neurosurgery. 1998 Jul;43(1):51-5. doi: 10.1097/00006123-199807000-00032. PMID 9657188

DOCUMENTS (1):
  • Informed Consent Form (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT03312192/ICF_000.pdf